CLINICAL TRIAL: NCT02498912
Title: A Phase I Clinical Trial of Cyclophosphamide Followed by Intravenous and Intraperitoneal Infusion of Autologous T Cells Genetically Engineered to Secrete IL-12 and to Target the MUC16ecto Antigen in Patients With Recurrent MUC16ecto+ Solid Tumors
Brief Title: Cyclophosphamide Followed by Intravenous and Intraperitoneal Infusion of Autologous T Cells Genetically Engineered to Secrete IL-12 and to Target the MUC16ecto Antigen in Patients With Recurrent MUC16ecto+ Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Stanford University (Other); Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-014
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors
Keywords: T Cells; Cyclophosphamide; MUC16ecto antigen; Intraperitoneal Infusion; Maximum Tolerated Dose (MTD); 15-014
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: This is a standard phase I dose escalation trial.

ARMS (1):
- Cyclophosphamide followed by Autologous T Cells (Experimental): Cohorts of 3-6 pts will be infused with escalating doses of modified T cells to establish the MTD of modified T cells. There are 5 planned dose levels: 3 x 10^5, 1 x 10^6, 3 x 10^6, & 1 x 10^7 & 3 x 10^7 4H11-28z/fIL-12/EGFRt+ T cells/kg. Cohort I-IV & VI will be treated escalating dose levels. Once the MTD of T cells is established, the next cohort will receive lymphodepleting cyclophosphamide dose of 750 mg/m^2 or a regimen of cyclophosphamide dose 300 mg/m2 x 3 days concurrent with fludarabine dose 25-30 mg/m2 x 3 days 2-7 days prior to starting the T cell infusion at one dose level below the MTD. If MTD isn't established after Cohort IV, Cohort V will receive conditioning chemotherapy 2-7 days prior to starting the T cell infusion at the same dose as Cohort III. Pts in Cohort V received cyclophosphamide chemotherapy on Day 1 or cyclophosphamide concurrent with fludarabine on Day 1-3, followed 2 to 4 days later by T cell infusion. This cohort is closed to further accrual.
  Interventions: Procedure: Production of Genetically-modified T cells; Drug: Cyclophosphamide; Device: IP Catheter Insertion; Genetic: Infusion of 4H11-28z/fIL-12/EGFRt+ Genetically-modified T cells; Drug: Fludarabine

INTERVENTIONS:
Procedure: Production of Genetically-modified T cells
Drug: Cyclophosphamide
Device: IP Catheter Insertion
Genetic: Infusion of 4H11-28z/fIL-12/EGFRt+ Genetically-modified T cells — Patients who do not have sufficient CAR T cells for the assigned dose cohort will be treated in the cohort for which cells are available.
Drug: Fludarabine — fludarabine dose 25-30 mg/m2 x 3 days

SUMMARY:
The purpose of this phase I study is to test the safety of different dose levels of specially prepared cells collected called "modified T cells". In the screening part of this study the tumor was found to have a protein called MUC16. This protein is present on about 70% of ovarian cancers. The investigators want to find a safe dose of modified T cells for patients with this type of cancer that has progressed after standard chemotherapy. We also want to find out what effects these modified T cells have on the patient and their cancer.

DETAILED DESCRIPTION:
There are 2 phases to the study: the Screening Phase and the Intervention Phase. Only patients identified as eligible from the Screening Phase may enroll in the Intervention Phase.

Screening Phase: After signing Informed Consent 1 (Screening Informed Consent), the patient's MUC16ecto tumor expression will be determined as previously described. In order to be eligible for this protocol, the patient's ovarian, primary peritoneal or fallopian tube carcinoma must express the MUC16ecto protein detectable by IHC analysis of banked (paraffin embedded) or fresh biopsied tumor. After signing Informed Consent 1, approximately 2 weeks will elapse while the patient's banked tumor is tested for MUC16ecto expression. If a patient's tumor is found to express MUC16ecto, she will undergo leukapheresis for the collection of peripheral blood mononuclear cells (PBMC), which will be frozen for future use. The leukapheresis product will be stored until the end of the study in case future research tests related to this study are developed.

Intervention Phase: Patients must sign Informed Consent 2 (Intervention Informed Consent) before receiving treatment on the study before receiving treatment on the study.

Once the patient is eligible to receive the CAR+ T cells, the frozen leukapheresis product will be thawed and used to generate the 4H11-28z/fIL-12/EGFRt+ genetically-modified T cells. It is expected to take approximately 4-6 weeks to prepare the autologous CAR+ T cells.

On day 1-3 patients in cohorts V will receive conditioning chemotherapy with cyclophosphamide 750 mg/m^2 or 300 mg/m2 cyclophosphamide concurrent with 25-30 mg/m2 fludarabine 2-7 days prior to the initial infusion of autologous CAR+T cells. Patients will receive autologous CAR+T cells in 2 infusions, the first IV and the second IP, each comprising about half the total dose. The IV infusion will be given first. The patient will then be closely monitored. One to 3 days later if clinically stable, the patient will receive the remaining dose of CAR+T cells IP. Patients in cohort I or -I will not receive cyclophosphamide, but will receive the T cells in the same manner (approximately half IV, followed by close monitoring and then 1-3 days later, if the patient is clinically stable, the remaining cells will be administered IP).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of high-grade serous ovarian, primary peritoneal, or fallopian tube carcinoma
* Presence of measurable recurrence, with RECIST measurable disease at the time of intervention consent
* Patient's carcinoma must express the MUC16ecto antigen detectable by IHC analysis of banked (paraffin embedded) or freshly biopsied tumor
* IHC evidence of MUC16ecto expression will be performed according to the technique and 0-5 scoring system described by Dharma et al (63)
* Only MUC16ecto tumors with moderate to strong immunoreactive scores (3-5) will be considered positive
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of ovarian, primary peritoneal, or fallopian tube carcinoma and at least two prior chemotherapy regimens.
* Patients are allowed to receive, but are not required to receive, up to 5 additional prior chemotherapy treatment regimens (including platinum-based chemotherapy). Prior hormonal therapy is allowed, does not count towards this prior regimen requirement, and must be discontinued at least one week prior to T cell infusion. Continuation of hormone replacement therapy is permitted
* Patients are allowed to receive, but are not required to receive, biologic/targeted therapy as part of their primary treatment regimen. Patients are allowed to receive, but are not required to receive, up to 5 biologic/targeted therapies as part of their treatment regimen for recurrent disease (either alone or in combination with chemotherapy)
* Karnofsky Performance Status score of 70% or greater
* Life expectancy of at least 3 months
* Adequate bone marrow, renal, and hepatic function:
* Absolute neutrophil count (ANC) ≥ 1500/mm³
* Platelets ≥ 100,000/mm³
* Creatinine ≤ 1.5mg/dL or creatinine clearance > 60ml/min
* ALT, AST, and total bilirubin all < 2.5 x the institutional upper limit of normal (ULN)
* Adequate pulmonary and cardiac function: No clinical evidence of cardiopulmonary disease, which, in the opinion of the investigator, precludes enrollment
* Age ≥18 years
* No anti-cancer therapy (chemotherapy, biologic therapy, or immunotherapy) in the 3 weeks prior to the T cell infusion (and all hematologic effects have resolved). No prior immunotherapy with checkpoint blockade (i.e. PD1 inhibitor, PDL1 inhibitor or CTL4-antagonist or similar agent) in the 6 months prior to the T cell infusion (and all clinically significant related side-effects related must be resolved).

Exclusion Criteria:

* Known active hepatitis B infection, known history of hepatitis C or HIV infection
* Clinical or radiographic evidence of bowel obstruction, or need for parenteral hydration and/or nutrition
* Known or suspected extensive abdominal adhesions.
* Any of the following cardiac conditions:
* Clinically significant heart disease (NYHA class III or IV) or symptomatic congestive heart failure
* Myocardial infarction ≤6 months prior to enrollment
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
* History of severe non-ischemic cardiomyopathy with ejection fraction ≤20%
* Active autoimmune disease (excluding autoimmune thyroid disease on a stable thyroid regimen). Such conditions include but are not limited to systemic lupus erythematous, rheumatoid arthritis, ulcerative colitis, Crohn's disease and temporal arteritis.
* Known or suspected leptomeningeal disease; patients with metastases to the brain stem, midbrain, pons or medulla.
* Known or suspected untreated brain metastases. Patients with Radiographically stable, asymptomatic previously irradiated lesions are eligible provided patient is ≥4weeks beyond completion of cranial irradiation and ≥ 3 weeks off of corticosteroid therapy at the time of study intervention.
* Prior history of seizure disorder
* Any concurrent active malignancies, defined as malignancies requiring any therapy other than expectant observation, since adverse events resulting from these malignancies or their treatment may confound our assessment of the safety of adoptive T cell therapy for ovarian cancer.
* Prior radiotherapy to any portion of the abdominal cavity or pelvis
* Current pregnancy or lactation
* Any of the following within 28 days of first date of study treatment:
* Serious uncontrolled medical illness or disorder that in the opinion of the treating physician would make the patient ineligible for the study
* Active uncontrolled infection (with the exception of uncomplicated urinary tract infection)
* Abdominal fistula, gastrointestinal perforation or intra-abdominal abscess
* Abdominal surgery (for reasons other than IP port placement)
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 2 years
  There are 5 planned dose levels of 4H11-28z/fIL-12/EGFRt+ T cells: 3 x 10^5, 1 x 10^6, 3 x 10^6, and 1 x10^7 and 3 x10^7 4H11-28z/fIL-12/EGFRt+ T cells/kg. The first subject will be treated at dose level 1 (3 x 10^5 4H11-28z/fIL-12/EGFRt+ T cells/kg). At least one week will elapse from the first patient's T cell infusions before the second patient is treated (on dose level 1) to allow for toxicity and safely assessment. 3 subjects will be enrolled in cohort I and followed for 30 days for safety assessments. If no DLT is observed after all three subjects have been observed for 30 days, a second cohort of 3 subjects will be enrolled at the same dose level (3 x 10^54H11-28z/fIL-12/EGFRt+ T cells/kg) with the addition of cyclophosphamide plus or minus fludarabine.

SECONDARY OUTCOMES:
evidence of anti-tumor activity | 2 years
  which will be defined according to the RECIST criteria, version 1.1 and, in appropriate subjects, the immune-related Response Criteria (irRC) (80)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin O'Cearbhaill, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/